CLINICAL TRIAL: NCT07033793
Title: Evaluation of a Preventive Intervention for Student Musicians, Independently Achievable, to Improve Good Health Behaviors: A Randomized Controlled Pilot and Feasibility Study.
Brief Title: Evaluation of the Effectiveness of Application-Supported Preventive Advice on Student Musicians' Health
Acronym: HarMoNie
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne-Violette Bruyneel (Other)
Collaborators: Geneva University of Music (Unknown)
Responsible Party: Sponsor-Investigator, Anne-Violette Bruyneel, Professor, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HarMoNie-129810; 2025-00300 (Other: Cantonal Commission for Ethics in Human Research (CCER))
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adults
Keywords: Prevention; Student musicians; Digital tool; Health knowledge

STUDY DESIGN:
Intervention Model Description: Number of Arms: 3
  * Preventive advice with digital support + educational sessions (GAppE)
  * Preventive advice with digital support only (GApp)
  * Control group with no intervention (GC)
Who Masked: Outcomes Assessor
Masking Description: Blinded, Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GC (No Intervention): Control group with no intervention.
- GApp (Experimental): Preventive advice with digital support
  Interventions: Behavioral: GApp
- GappE (Experimental): Preventive advice with digital support + 5 educational sessions
  Interventions: Behavioral: GappE

INTERVENTIONS:
Behavioral: GApp — Participants receive only digital support with health information, self-assessment tests, preventive advices and games. No educational sessions are provided, and the focus is solely on digital preventive advice used autonomously.
  Arms: GApp
Behavioral: GappE — Participants receive preventive interventon delivered via digital support (smartphone app) including health information, self-assessment tests, preventive advices and games).
  In addition to the App used autonomously, they will participate in 5 group educational sessions proposed by a physiotherapist (once every two weeks).
  Arms: GappE

SUMMARY:
Student musicians are particularly vulnerable to both physical and psychological health issues, with studies showing that 38% report pain from musical practice and over 50% experience high stress. Despite these risks, health resources tailored specifically to student musicians remain limited. This study aims to address this gap by testing a preventive, digital intervention to improve the well-being of this population. The intervention, delivered via a smartphone or tablet app, is designed to accommodate the unique demands of student musicians, such as frequent travel and time constraints. It includes health education, self-assessment tools, preventive health behavior advice, and interactive games designed to promote healthier work habits, daily routines, and overall health knowledge.

DETAILED DESCRIPTION:
Student musicians are significantly affected by physical and psychological health issues. Previous studies highlighted that 38% of student musicians experience pain related to their musical practice over a 12-month period, and more than 50% report high levels of stress (general and specific to musical performance).

Despite these concerning trends, tailored health resources and advice specific to student musicians remain rare. Improved work habits and daily health behaviors are crucial for primary prevention and could enhance both learning conditions and long-term health despite the high level of musical practice. Digital, evidence-based interventions, tailored to the specific needs of musicians, could offer a practical solution given their unique constraints, which include frequent travel, limited resources, and demanding schedules.

This study aims to evaluate the feasibility and effectiveness of a smartphone/tablet-based preventive intervention for student musicians. The intervention is designed to improve their physical, psychological, and social well-being, as well as health knowledge. Given the health risks associated with pre-professional and professional music practice, these issues impact not only the well-being of student musicians but also their self-fulfillment and learning capacity. These issues justify the need for health support in music studies. It is currently recommended to develop health promotion approaches that integrate knowledge about health, self-assessment of risk factors, and the adoption of good daily habits. These approaches are most effective when tailored to the specific needs of musicians.

This study will assess a preventive, digital intervention for student musicians over a 12-week period. The three groups involved are: GAppE (stand-alone app intervention plus 5 educational group sessions), GApp (app intervention used independently), and GC (no intervention).

Health knowledge, physical, psychological, and social well-being, as well as daily life and work habits, will be assessed at three time points: 1) before the intervention, 2) 6 months after the start of the intervention, and 3) 12 weeks after the start of the intervention in all 3 groups.

Moreover, after 6 and 12 weeks, participants in the GAppE and GApp groups will also evaluate their satisfaction with the app-based preventive intervention using standardized questionnaires.

The hypothesis is that the intervention will be feasible, useful, and appreciated, and that it will have beneficial health outcomes, particularly when combined with educational group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18 years old
* Enrollment at the Geneva University of Music (HEM) as a Bachelor (1st, 2nd, or 3rd year) or Master (1st or 2nd year) student.
* Primary discipline: Must be in musical performance (instrumental or vocal).
* Physical ability to play an instrument or sing (no physical disabilities that prevent participation in musical practice).
* Must be able to follow academic activities as planned.

Exclusion Criteria:

* Unable to play their instrument or participate in singing.
* Underwent surgery in the past 12 months that affects their ability to practice music (e.g., musculoskeletal surgeries).
* Suffering from pain or medical conditions that are not related to musical practice (e.g., non-musical injuries or pathologies).
* Unable to follow the planned academic schedule (e.g., missing classes or major academic constraints that would prevent full participation in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Participant Interest in the App-Based Intervention | At baseline.
  As part of the feasibility assessment guided by the CONSORT extension for pilot and feasibility trials, this outcome evaluates the attractiveness of the application-based intervention, measured by the number of participants who will express interest in the intervention at baseline.
Participant Engagement with and Frequency of Use of the App - Based Intervention | From the start of the intervention to 12 weeks.
  This outcome measures the use of the app-based intervention as part of the feasibility assessment. Use is evaluated by tracking the frequency of mobile app access by each participant throughout the intervention period.
Participant Satisfaction with the App-Based Intervention | 6 and 12 weeks after the start of intervention.
  Participant satisfaction is measured using a Visual Analog Scale (VAS), where participants rate their overall satisfaction from 0 (not satisfied) to 10 (fully satisfied).
System Usability of the App-Based Intervention Using SUS | 6 and 12 weeks after the start of intervention.
  This outcome assesses the usability of the mobile app-based intervention using the System Usability Scale (SUS), which is a validated 10-item questionnaire designed to evaluate perceived ease of use. The total SUS score ranges from 0 to 100, with higher scores indicating better perceived usability. This measure is part of the feasibility assessment guided by the CONSORT extension for pilot and feasibility trials.
Participant Satisfaction with the App-Based Intervention | 6 and 12 weeks after the start of intervention.
  As part of the feasibility assessment guided by the CONSORT extension for pilot and feasibility trials, this outcome evaluates participant satisfaction with the mobile app using the Visual Analog Scale (VAS): satisfaction scores at 6 and 12 weeks, where participants rate overall satisfaction from 0 (not satisfied) to 10 (fully satisfied).

SECONDARY OUTCOMES:
Assessment of the prevalence of Playing-related Muscoskeletal Disorders by using the Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians (MPIIQM). | Baseline, 6 weeks, 12 weeks after start of intervention
  This questionnaire is considered the gold standard for assessing musculoskeletal pain and discomfort related to practice of music. It evaluates the intensity of pain and its interference with musical performance with 22-items (8 for musician characteristics and 14 related with pain related with musical practice). The MPIIQM includes a subscale about pain intensity (0 to 40) and pain interference (0 to 50).
  Higher scores indicate greater pain intensity and interference with musical practice.
Change in Health-Related Quality of Life as Measured by the SF-36 Health Survey | Baseline, 6 weeks, 12 weeks after start of intervention
  The SF-36 assesses the perceived physical and mental quality of life across eight dimensions: physical functionning (10 items), role limitations (4 items); bodily pain (2 items); general health perceptions (5 items); energy/vitality (4 items); social functioning (2 items); emotional role limitations (3 items); general mental health (5 items) and health transition (1 item). The total score ranges from 0 to 30. Higher score indicates better perceived health-related quality of life.
Change in Psychosocial Adaptation Scores on the Health Interview for Musicians (HIL) Scale | Baseline, 6 weeks, 12 weeks after start of intervention
  The questionnaire assesses professional health and psychosocial adaptation among musicians. It evaluates multiple dimensions relevant to musical performance, including 7 domains: satisfaction with professional achievement, confidence in stage situations, breathing while playing, satisfaction with posture, movement sensations, symptoms during performance, and perceived ability to meet musical demands. The total score ranges from 6 to 42. High score shows good adaptability to constraint. Changes in this score may reflect the impact of the preventive intervention on physical and mental health in the context of musical work.
Change in Psychological Distress Scores on the Kessler Psychological Distress Scale (K10) | Baseline, 6 weeks, 12 weeks after start of intervention
  The Kessler Psychological Distress Scale (K10) is a validated 10-item self-report questionnaire designed to assess symptoms of anxiety and depression over the past 4 weeks. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low score indicates low levels of psychological distress and high scores indicate high levels of psychological distress. Since student musicians have a high level of general stress, a change will allow us to observe whether interventions have an effect on this risk factor.
Change in Music Performance Anxiety Scores on the Kenny Music Performance Anxiety Inventory (K-MPAI-R) | Baseline, 6 weeks, 12 weeks after start of intervention
  The K-MPAI-R is a validated 40-item with a 7-point Likert scale measuring anxiety related to music performance specific to the target population. Total score: 7 to 280 points. A high total score corresponds to high anxiety and distress regarding musical performance and vice versa. Since student musicians have a high level of performance-related stress, a change will allow us to observe whether interventions have an effect on this risk factor.
General Fatigue Rating | Baseline, 6 weeks, 12 weeks after the start of the intervention.
  Following recommendations from a Delphi consensus study, a general fatigue rating is collected. Participants rate their current level of fatigue using a single-item self-report scale ranging from 0 (no fatigue) to 10 (maximum fatigue), providing a quick global indicator of perceived fatigue.
Fatigue Change and Recovery as Measured by the McCrary Fatigue Scale | Baseline, 6 weeks, 12 weeks after the start of the intervention.
  Fatigue will also be assessed using the McCrary Fatigue Questionnaire. It is a 5-item validated scale developed specifically for musicians. It evaluates dimensions such as pain, sleep, recovery, workload, and physical condition. Items are rated on a 0-10 scale. A high total score represents greater fatigue. The intervention includes education on fatigue management, which may impact both perceived and reported fatigue levels.
Occupational Balance as Measured by OBQ | Baseline, 6 weeks, 12 weeks after start of intervention
  The Occupational Balance Questionnaire (OBQ) is used to evaluate satisfaction with how time is spent and the variety of activities undertaken. A 13-item self-report scale. Each item is scored 0-3; total score range: 0-39. Higher score represents better occupational balance.The advice includes recommendations for time management, periodization, and health-promoting activities. A change will highlight whether the interventions have an effect on occupational balance.
Change in Musicians' Health Literacy Scores Measured by the MHL-Q19 Questionnaire | Baseline, 6 weeks, 12 weeks after start of intervention
  Health literacy will be assessed using the Musicians' Health Literacy Questionnaire (MHL-Q19), a 19-item scale developed specifically for student musicians. It evaluates the ability to access, understand, and apply health information across clinical care, prevention, and health promotion contexts. Each item is scored as either difficult (0) or easy (1), producing a total score ranging from 0 to 19. Scores are categorized as:
  * Inadequate (0-9)
  * Problematic (10-14)
  * Sufficient (15-19). The app includes information on health and good behaviors. A change will highlight the effects on health knowledge.
Change in the Self-Perceived Musical Performance Quality Assessed by a Visual Analog Scale | Baseline, 6 weeks, 12 weeks after start of intervention
  Self-perceived performance quality will be measured using a Visual Analog Scale (VAS) ranging from 0 (lowest imaginable performance) to 10 (best imaginable performance). Participants will rate their average performance quality over the previous 3 days. This outcome assesses the participant's subjective perception of their musical performance and whether it is influenced by the preventive intervention.
General Self-Efficacy (GSES) | Baseline, 6 weeks, 12 weeks after start of intervention
  The General Self-Efficacy Scale (GSES) assesses confidence in one's coping ability in difficult situations with 10-items. Each item is evaluated with a 4-point scale (1 = not at all true and 4 = absolutely true). The total score ranges from 10 to 40. Higher scores reflect stronger self-efficacy.

OTHER OUTCOMES:
Demographic Information at Baseline | Baseline (pre-intervention)
  Baseline demographic data will be collected, including age, sex, type of musical discipline background, general health history, prior musculoskeletal pain or disorders (PRMDs), any other extracurricular activities outside of music studies, work and music practice habits, and lifestyle habits. This information will be used to characterize the study sample and explore potential demographic and baseline factors that may influence study outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva School of Health (HEdS-Geneva), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures may be provided to qualified researchers. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after the study completion and after the major publications have been submitted
Access Criteria: At the end of the project, the data will be deposited in repository developed by the University of Geneva. This choice will ensure that data is archived and shared in accordance with FAIR principles.

REFERENCES:
- [Background] Bruyneel AV, Stern F, Schmid A, Rieben N, James CE. Network analyses of physical and psychological factors of playing-related musculoskeletal disorders in student musicians: a cross-sectional study. BMC Musculoskelet Disord. 2024 Nov 30;25(1):979. doi: 10.1186/s12891-024-08103-8. PMID 39616356